CLINICAL TRIAL: NCT02673840
Title: Ketotifen as a Treatment for Vascular Leakage During Dengue Fever (KETODEN)
Brief Title: Ketotifen as a Treatment for Vascular Leakage During Dengue Fever
Acronym: KETODEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EID-DF-02
Record Dates: First submitted 2015-10-30; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Dengue Fever; Pleural Effusion
Keywords: dengue fever; dengue hemorrhagic fever; ketotifen; vascular leakage; pleural effusion; plasma leakage
MeSH Terms: conditions — Dengue; Pleural Effusion; Severe Dengue | interventions — Ketotifen; ketotifen fumarate ophthalmic solution; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketotifen (Experimental)
  Interventions: Drug: Ketotifen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketotifen — 2 mg of Ketotifen, twice a day for a total of ten (10) doses
  Other Names: Zaditor; C19H19NOS; Drugbank Identifier: DB00920
  Arms: Ketotifen
Drug: Placebo — Identical tablets containing 0 mg of Ketotifen, twice a day for a total of ten (10) doses
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Rationale and Aims: Infection by dengue virus (DENV) causes major morbidity and mortality throughout the world. In 2012, an estimated 3.6 billion people live in areas at risk for DENV infection, including Singapore. The key pathology of DENV infection is vascular leakage, which can occur in mild cases and can become life-threatening in severe cases when patients may develop dengue hemorrhagic fever (DHF) or dengue shock syndrome (DSS). Mast cells (MCs) are strongly activated by DENV with preliminary studies showing that activation levels are correlated to disease severity in human patients. Thus, the investigators propose to use the MC stabilizing drug, ketotifen, to limit the immune pathology that is characteristic of dengue infection and treat dengue-induced vascular leakage. Methods: The ability of Ketotifen to reduce vascular leakage in DENV patients will be determined by assessing the pooling of fluid in the pleural cavity (measured by MRI and CXR) after 5 days of drug administration, evaluated as a percent change compared to baseline fluid levels. Additional measures of vascular leakage and immune pathology will be compared as secondary objectives. The trial will be conducted as a randomized, double-blind study comparing the responses of dengue patients given either ketotifen or placebo (n=55 per arm). Importance of proposed research: Currently, no targeted treatments exist to limit vascular leakage during DENV infection. If Ketotifen is identified as effective for preventing pleural effusion and/or plasma leakage in DENV patients, this would constitute an advance for the clinical management of DENV fever. This finding would also support a large-scale trial to determine whether Ketotifen can be used to prevent severe vascular leakage as occurs during DHF/DSS. Benefits/Risks: Ketotifen has a record of safety and tolerability in humans, regulatory approval, and widespread use. Side effects are generally mild. The potential exists that, if effective, many of the painful and life-threatening symptoms of DENV infection that result from plasma leakage would be improved.

DETAILED DESCRIPTION:
Approximately 230 million individuals are infected each year by dengue virus (DENV) a Flavivirus spread by mosquito vectors that causes substantial worldwide morbidity and mortality. Infection by DENV results in dengue fever (DF), which is usually a self-limiting illness. However, many individuals can experience much more severe forms of disease, such as dengue hemorrhagic fever (DHF) and dengue shock syndrome (DSS), which are characterized by widespread vascular pathology, the most prominent manifestation of which is plasma leakage that can lead to shock and, potentially, death. Currently, treatment for DHF/DSS is supportive care with analgesics, fluid replacement and bed rest. Management of severe DENV infections typically requires prolonged hospitalization accompanied by careful fluid management . At this time, there are no targeted treatments for DF, DHF or DSS, making improvements in care for DENV patients an urgent clinical need. In particular, there is a need for therapeutic intervention to prevent the vascular leakage.

Animal studies suggested that drugs in the class of mast cell (MC) "stabilizers" can effectively limit vascular leakage in mouse models of DENV infection. Drugs targeting MCs have been in use in humans for decades, particularly for the treatment of allergy and asthma. One "MC stabilizer", ketotifen, acts by preventing degranulation of MCs. Ketotifen is an oral drug currently used to prevent asthma. It is most commonly supplied in the form of a salt with fumaric acid, as ketotifen fumarate. Ketotifen has a clinical track record of greater than 30 years as a safe drug and it is currently approved for use in Singapore. In other formulations it is also used to treat irritation and reduce vascular leakage, such as in the eye. It is a MC stabilizing agent that prevents degranulation of MCs, as well as the production of additional mediators that are not contained within MC granules, including leukotrienes and platelet activating factor. Ketotifen also functions as an antihistamine with direct H1-receptor blocking function. The bioavailability of an oral dose of ketotifen in humans is approximately 80-90% . Drug levels peak in the serum between 2-4 hours after ingestion. Patients with asthma sometimes require treatment with ketotifen for weeks prior to observing improved asthmatic responses, but this is thought to represent the time required for chronic inflammation to subside and not the time required for MC stabilization, which occurs immediately in animal models. The mean elimination half-life of ketotifen is 12 hours. Side effects include drowsiness, dry mouth, slight dizziness, central nervous system (CNS) stimulation and weight gain. Patients are commonly prescribed 1-2mg tablets, twice a day. Treatment of DENV-infected mice with MC stabilizers, cromolyn or ketotifen, resulted reduced vascular leakage compared to untreated controls in two separate mouse models of DENV infection. These findings were apparent using two separate measures of vascular leakage as the endpoint readout: evans blue perfusion, which is a key experimental technique to show plasma leakage into tissues, and hematocrit analysis, which is the clinical parameter that is most commonly used to diagnose DHF in human patients.

This is a randomized, double blind, placebo-controlled, clinical study of ketotifen in adults with dengue infection. The study will be conducted as an outpatient study at National University Hospital (NUH) and Singapore General Hospital (SGH), daily with the MRIs and chest X-rays conducted at the Clinical Imaging Research Centre (CIRC) of the National University of Singapore (NUS). A final visit at convalescence (Day 21) can be at the site of enrolment. One hundred and ten (110) patients will be randomized 1:1 to ketotifen or placebo. A baseline MRI of the pleural cavity, liver, spleen and kidney will be taken. Tablets of placebo or ketotifen will be self-administered for 5 days. Patients will be given daily clinical exams, Day 1 to Day 5, and blood samples will be collected for plasma chymase levels, viral load, hematology, clinical chemistry, inflammatory product profiling and additional laboratory tests. After the administration of the final dose of drug, blood will be drawn and a follow up MRI will be performed at the CIRC in NUS to assess fluid accumulation within the pleural cavity as a primary clinical endpoint, with assessment of the liver, spleen and kidney as experimental endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 21-60 years
2. Fever of ≥ 37.5°C (directly measured or patient reported) of ≤ 72 hr duration.
3. Positive Nonstructural protein 1 (NS1) strip assay or dengue polymerase chain reaction (PCR)
4. Able and willing to give written or oral informed consent
5. Willing to be an outpatient from Study Day 1 to 5, to undergo an MRI and chest X-ray day 1 at the hospital, to return to the hospital on day 5 for an MRI and chest X-ray, and return on Study Days 7 and 21.
6. Willing to keep a diary of pain medication usage and side effects

Exclusion Criteria:

1. Clinical signs and symptoms for severe dengue, such as: a. Persistent vomiting b. Altered mental state c. Liver enlargement > 2 cm
2. A person with any of the following laboratory values: a. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 1000 U/L
3. Current usage of any anticoagulant drugs including, but not limited to, aspirin, warfarin, or clopidogrel.
4. Current usage of any drugs that are known to block the functions of ketotifen, such as propranolol.
5. Current usage of oral anti-diabetic agents.
6. Any other clinically significant acute illness within 7 days prior to first study drug administration.
7. Patients with renal impairment.
8. Exposure to any new investigational agent within 30 days prior to the study drug administration.
9. Clinically significant abnormal physical examination unrelated to dengue infection.
10. Females of childbearing potential who are pregnant, breast feeding, or unwilling to avoid pregnancy by the use of appropriate contraception, including oral and subcutaneous implantable hormonal contraceptives, condoms, diaphragm, or intrauterine device (IUD), during the period that the experimental drug is administered. Prospective female participants of childbearing potential must have a negative pregnancy test (point of care).
11. Current significant medical condition or illness including cardiac arrhythmias, cardiomyopathy or other cardiac disease, immunocompromised state including known HIV infection, or any other illness that the Investigator considers should exclude the patient, especially those that require continuation of other medications likely to have an interaction with the study drug. Patients with a history of allergy will not be excluded unless the allergy may be directed to the Study Drug or other tablet ingredient.
12. Any condition that would render the informed consent invalid, or limit the ability of the patient to comply with the study requirements.
13. Any condition that, in the opinion of the investigator, would complicate or compromise the study or well being of the patient.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
reduced fluid accumulation in the pleural cavity | day 5-7
  fluid accumulation in the pleural cavity will be measured by MRI

SECONDARY OUTCOMES:
reduced serum biomarker chymase | day 5-7
  Serum biomarker for mast cell activation, chymase, will be measured in serum
reduced hemoconcentration | day 5-7
  hemoconcentration will be measured by hematocrit
Number of patients with symptoms associated with DF | day 5-7
  This is determined by the presence of rash, petechiae, purpura, ecchymoses, epistaxis, or other signs of bleeding, pain, or discomfort
time to viral clearance | day 5-7

OTHER OUTCOMES:
Number of patients with abnormal immunoprofiles | day 5-7
  Factors taken into account include: RNA expression levels, plasma chymase levels, viral load, hematology (full blood count), viral protein levels, inflammatory cytokines, inflammatory lipids (such as eicosanoids), and expression of activation markers, and genetic factors
patients with Fluid accumulation in the liver, spleen or kidney | day 5-7
  fluid accumulation in the liver, spleen or kidney will be measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ashley L St John, Study Director — Duke-NUS Graduate Medical School; Paul A Tambyah, Principal Investigator — National University Hospital; National University of Singapore
Locations (2):
- Singapore (2):
  - National University Hospital (Investigational Medicine Unit), Singapore
  - Singapore General Hospital, Singapore

REFERENCES:
- [Background] St John AL, Rathore AP, Raghavan B, Ng ML, Abraham SN. Contributions of mast cells and vasoactive products, leukotrienes and chymase, to dengue virus-induced vascular leakage. Elife. 2013 Apr 30;2:e00481. doi: 10.7554/eLife.00481. PMID 23638300
- [Background] Syenina A, Jagaraj CJ, Aman SA, Sridharan A, St John AL. Dengue vascular leakage is augmented by mast cell degranulation mediated by immunoglobulin Fcgamma receptors. Elife. 2015 Mar 18;4:e05291. doi: 10.7554/eLife.05291. PMID 25783751
- [Background] Dengue: Guidelines for Diagnosis, Treatment, Prevention and Control: New Edition. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK143157/ PMID 23762963
- [Background] Halstead SB. Dengue. Lancet. 2007 Nov 10;370(9599):1644-52. doi: 10.1016/S0140-6736(07)61687-0. PMID 17993365
- [Background] Craps LP. Immunologic and therapeutic aspects of ketotifen. J Allergy Clin Immunol. 1985 Aug;76(2 Pt 2):389-93. doi: 10.1016/0091-6749(85)90659-1. PMID 4019961
- [Background] Disodium cromoglycate. Lancet. 1972 Dec 16;2(7790):1299. No abstract available. PMID 4117822
- [Background] Abraham SN, St John AL. Mast cell-orchestrated immunity to pathogens. Nat Rev Immunol. 2010 Jun;10(6):440-52. doi: 10.1038/nri2782. PMID 20498670
- [Background] Atrasheuskaya A, Petzelbauer P, Fredeking TM, Ignatyev G. Anti-TNF antibody treatment reduces mortality in experimental dengue virus infection. FEMS Immunol Med Microbiol. 2003 Jan 21;35(1):33-42. doi: 10.1111/j.1574-695X.2003.tb00646.x. PMID 12589955
- [Background] Gowen BB, Julander JG, London NR, Wong MH, Larson D, Morrey JD, Li DY, Bray M. Assessing changes in vascular permeability in a hamster model of viral hemorrhagic fever. Virol J. 2010 Sep 16;7:240. doi: 10.1186/1743-422X-7-240. PMID 20846417
- [Background] Humbert H, Cabiac MD, Bosshardt H. In vitro-in vivo correlation of a modified-release oral form of ketotifen: in vitro dissolution rate specification. J Pharm Sci. 1994 Feb;83(2):131-6. doi: 10.1002/jps.2600830205. PMID 8169778
- [Background] Kunder CA, St John AL, Abraham SN. Mast cell modulation of the vascular and lymphatic endothelium. Blood. 2011 Nov 17;118(20):5383-93. doi: 10.1182/blood-2011-07-358432. Epub 2011 Sep 8. PMID 21908429
- [Background] McClean SP, Arreaza EE, Lett-Brown MA, Grant JA. Refractory cholinergic urticaria successfully treated with ketotifen. J Allergy Clin Immunol. 1989 Apr;83(4):738-41. doi: 10.1016/0091-6749(89)90008-0. PMID 2651507
- [Background] Oliveira GA, Machado RC, Horvat JV, Gomes LE, Guerra LR, Vandesteen L, Oliveira FT, Lousada NS, Moreira-Silva S, de Fatima Ceolin M. Transient reticular gallbladder wall thickening in severe dengue fever: a reliable sign of plasma leakage. Pediatr Radiol. 2010 May;40(5):720-4. doi: 10.1007/s00247-009-1489-x. Epub 2009 Dec 15. PMID 20012951
- [Background] Sendo T, Sumimura T, Itoh Y, Goromaru T, Aki K, Yano T, Oike M, Ito Y, Mori S, Nishibori M, Oishi R. Involvement of proteinase-activated receptor-2 in mast cell tryptase-induced barrier dysfunction in bovine aortic endothelial cells. Cell Signal. 2003 Aug;15(8):773-81. doi: 10.1016/s0898-6568(03)00014-7. PMID 12781870
- [Background] St John AL, Rathore AP, Yap H, Ng ML, Metcalfe DD, Vasudevan SG, Abraham SN. Immune surveillance by mast cells during dengue infection promotes natural killer (NK) and NKT-cell recruitment and viral clearance. Proc Natl Acad Sci U S A. 2011 May 31;108(22):9190-5. doi: 10.1073/pnas.1105079108. Epub 2011 May 16. PMID 21576486
- [Background] Theoharides TC, Sieghart W, Greengard P, Douglas WW. Antiallergic drug cromolyn may inhibit histamine secretion by regulating phosphorylation of a mast cell protein. Science. 1980 Jan 4;207(4426):80-2. doi: 10.1126/science.6153130.
- [Background] Venkata Sai PM, Dev B, Krishnan R. Role of ultrasound in dengue fever. Br J Radiol. 2005 May;78(929):416-8. doi: 10.1259/bjr/54704044. PMID 15845934
- [Background] Wilder-Smith A, Renhorn KE, Tissera H, Abu Bakar S, Alphey L, Kittayapong P, Lindsay S, Logan J, Hatz C, Reiter P, Rocklov J, Byass P, Louis VR, Tozan Y, Massad E, Tenorio A, Lagneau C, L'Ambert G, Brooks D, Wegerdt J, Gubler D. DengueTools: innovative tools and strategies for the surveillance and control of dengue. Glob Health Action. 2012;5. doi: 10.3402/gha.v5i0.17273. Epub 2012 Mar 22. PMID 22451836